CLINICAL TRIAL: NCT04634097
Title: DECLIC Patient Education Program : Assessment Through a Population Health Intervention Research Approach (LE DECLIC EPRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IC 2019-06
Record Dates: First submitted 2020-10-30; First posted 2020-11-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Cancer Patients With Cancer Pain

STUDY DESIGN:
Intervention Model Description: Control group : Standard follow-up patient related to pain. Specific to each center : with or without existing local ETP program (standard care).
  Experimental group : Clusters will be proposed LE DECLIC EPRI intervention, which is a complex intervention, associating 3 components,:
  A. DECLIC program set up in the centers, open to concerned patients.
  B. 3 training sessions :
  * one public of primary care physicians in order to give them the opportunity to be involved in the medical care in charge of the patient suffering from cancer pain.
  * one public of cancer physicians, leaders of opinions in each cancer centers participating to the study and one public of health professionals in order to train them to be educators (team building).
  * for healthcare professionals in order to train them as educators in this program.
  C. The collaboration of one primary care network, specialized in pain management, in order to reinforce the patient care pathway.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Clusters will be proposed LE DECLIC EPRI intervention, which is a complex intervention, associating 3 components,:
  A. DECLIC program set up in the centers, open to concerned patients.
  B. 3 training sessions :
  * one public of primary care physicians in order to give them the opportunity to be involved in the medical care in charge of the patient suffering from cancer pain.
  * one public of cancer physicians, leaders of opinions in each cancer centers participating to the study and one public of health professionals in order to train them to be educators (team building).
  * for healthcare professionals in order to train them as educators in this program.
  C. The collaboration of one primary care network, specialized in pain management, in order to reinforce the patient care pathway.
  Interventions: Other: Experimental group
- Standard group (Other): Standard follow-up patient related to pain. Specific to each center : with or without existing local ETP program (standard care).
  Interventions: Other: standrad group

INTERVENTIONS:
Other: Experimental group — Clusters will be proposed LE DECLIC EPRI intervention, which is a complex intervention, associating 3 components,:
  A. DECLIC program set up in the centers, open to concerned patients.
  B. 3 training sessions :
  * one public of primary care physicians in order to give them the opportunity to be involved in the medical care in charge of the patient suffering from cancer pain.
  * one public of cancer physicians, leaders of opinions in each cancer centers participating to the study and one public of health professionals in order to train them to be educators (team building).
  * for healthcare professionals in order to train them as educators in this program.
  C. The collaboration of one primary care network, specialized in pain management, in order to reinforce the patient care pathway.
  Arms: Experimental group
Other: standrad group — Standard follow-up patient related to pain. Specific to each center : with or without existing local ETP program (standard care).
  Arms: Standard group

SUMMARY:
Cancer pain is a frequent symptom, reported by 20 to 70% of patients in any stage of the cancer disease : 60 to 70% in the advanced stage of the disease and 20 to 40% among the survivors. Among patients who report pain, 40% report undertreated pain. Strengthening Pain management in cancer is a specific objective of the French Cancer Plan. Providing patient education for cancer pain management is recommended since small to moderate efficacy of patient education on pain intensity and interference was found in all meta-analysis. An effect size comparable with some analgesic agents. However, recommendations suggest improvement in order to increase effectiveness and population reach of those interventions. The DECLIC EPRI intervention aim at addressing all the issues raised by patient education for cancer pain management. It was developed according to the framework of Michie's Behavior change wheel theory.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged over 18.
2. Followed in the participant comprehensive cancer center.
3. All cancer types, location and stage.
4. Patient under any anticancer treatment (including hormonal therapy) or patient has stopped his treatment (including hormonal therapy) maximum 2 years before inclusion.
5. Patient experiencing cancer pain and/or his treatments for 3 months or more.
6. All previous and concomitant treatments are accepted.
7. Participation to another clinical trial is accepted.
8. Patient has accepted to participate to the study and signed informed consent form or his legal representative.
9. Patient affiliated to the social security healthcare.

Exclusion Criteria:

1. Cognitive impairment preventing to understand the patient education program.
2. Language barrier preventing to understand the patient education program.
3. Physical impairment preventing patient to attend to the patient education program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Effectiveness of LE DECLIC EPRI intervention on the pain interference with the daily life | 6 months
  Brief pain Inventory BPI Questionnaire

SECONDARY OUTCOMES:
Effectiveness of the intervention on other clinical outcomes | 6 months
  Brief pain Inventory BPI, EQ-5D, DAMS questionnaires Other dimension of the QCD : current pain, average pain and worst pain in the last 24 hours.
  Number of area identified as painfull by the patient, and surface of those area, measured on the "figures" item of the QCD.
  Quality of life, assessed with the EQ-5D, in order to transform the results into utilities for the efficiency evaluation.
  Side effects occurrence, related to the toxicity of the analgesics, assessed with a questionnaire constructed by the research team (questionnaires ad hoc).
  Occurrence of atypical pain. Date of the occurrence of atypical pain. Occurrence of epiduritis. Date of the occurrence of epiduritis. Time between atypical pain occurrence and epiduritis diagnosis. Adhesion to analgesic medications assessed with a French translation of the questionnaire DAMS (Garfield et al), standardized per analgesic.
The organizational effectiveness of the intervention. | 6 months
  Organizational effectiveness Number of GPs recruited in the training sessions. Number of other primary care professionals recruited in the training sessions. Number of consultations with the GP by patient. Number of cancer pain consultations with the GP by patient. Number of consultation by patient due to pain with the GP. Number of interactions developed between the pain management network and GPs. Number of emergency consultations and hospitalisations due to pain by patient in the center.
Educational effectiveness of the intervention. | 6 months
  quiz with certitude level assessement, sure test, HADS questionnaires, French-Canadian Chronic Pain Self-efficacy Scale (FC-CPSES).
  Knowledge, assessed with a quiz with certitude level assessement, developed specifically for the DECLIC program, by a multidisciplinary team of physicians, patients and reseachers.
  Skills assessed with scenarii (simulated cases) developed specifically for the DECLIC program, by a multidisciplinary team of physicians, patients and reseachers. Informed decision assessed with a scenario (simulated case) developed specifically for the DECLIC program, by a multidisciplinary team of physicians, patients and reseachers. Informed decision is assessed with the French version of the SURE test. Anxiety : with the HADS questionnaire. Self efficacy, with French-Canadian Chronic Pain Self-efficacy Scale (FC-CPSES).
  Sense of control with visual analogical scale. Ability to communicate with visual analogical scale developed specifically for the DECLIC program.
Effectiveness of the intervention on patients value. | 6 months
  D'Ivernois 2008 questionnaire, PAT-SAT 32 questionnaire, SMD Q9 questionnaire. Patient perceived quality of care will be assessed thanks to the medical consultation dimension of the PAT-SAT 32, a validated questionnaire in French.
  Reported share decision making, inside GPs consultation, by patient. Share decision making assessed in the center with the with the SMD Q9, validated in French.
Efficiency of the intervention. | 6 months
  Cost-effectiveness analysis.
Effect of patient's caracteristics on the intervention effectiveness and participation. | 6 months
  EDI quintile and Newest Vital Sign
Implementation of the intervention | 48 months
  participation rate in the training of GPs and KLOs, number of GPs contacting the network, number of GPs contacting the patient education team, number of oncologists referring patients to the DECLIC program, number of patients referred by oncologist, number of oncologist consulting the patient education DECLIC e-record.
  Reach :
  number of patients who agreed to participate/number of patients to whom the study was proposed.
  Reasons for refusal.
Interaction between the contexts and the intervention effectiveness. | 48 months
  Barriers and drivers to intervention adoption among KLOs and oncologists. Barriers and drivers to effective intervention in GPs. Barriers and drivers to effective intervention in patients.
Mechanisms of action of the intervention. | 48 months
  Unexpected outcomes.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Institut de Cancérologie de l'Ouest Paul Papin, Angers
  - Institut Curie, Paris
  - GH Diaconesses Croix Saint Simon (GHDCSS), Paris
  - AP-HP La Pitié Salpêtrière, Paris
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).